CLINICAL TRIAL: NCT05153486
Title: A Randomized Control Study of Catheter Ablation Versus Surgical Ablation as a Treatment in Patients With Persistent Atrial Fibrillation With Severe Atrial Fibrosis: a Chinese Registry Study.
Brief Title: Catheter Ablation and Surgical Ablation of Persistent Atrial Fibrillation With Severe Atrial Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAAF II
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; severe atrial fibrosis; catheter ablation; surgical ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation
  Interventions: Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation
- Group B (Active Comparator): Circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion
  Interventions: Procedure: Circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion
- Group C (Active Comparator): Surgical ablation
  Interventions: Procedure: Surgical ablation

INTERVENTIONS:
Procedure: Circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation — Patients receive circumferential pulmonary vein isolation and linear ablation (ablation of a roof line and a mitral isthmus line) combined with bi-atrial mapping and driver ablation.
  Arms: Group A
Procedure: Circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion — Patients receive circumferential pulmonary vein isolation and linear ablation (ablation of a roof line and a mitral isthmus line) combined with vein of Marshall ethanol infusion.
  Arms: Group B
Procedure: Surgical ablation — Patients receive surgical ablation.
  Arms: Group C

SUMMARY:
This is an open label, randomized parallel control clinical trial evaluating the efficacy and safety of catheter ablation and surgical ablation in patients with persistent atrial fibrillation with severe atrial fibrosis.

DETAILED DESCRIPTION:
This is an open label, randomized parallel control clinical trial. Patients with persistent atrial fibrillation with severe atrial fibrosis are 1:1:1 randomized into the group A (circumferential pulmonary vein isolation + linear ablation + bi-atrial mapping + driver ablation), group B (circumferential pulmonary vein isolation + linear ablation + vein of Marshall ethanol infusion) and group C (surgical ablation). Postoperative recurrence rate and other indicators are analyzed to evaluate the efficacy and safety of catheter ablation and surgical ablation in patients with persistent atrial fibrillation with severe atrial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old;
2. Persistent AF with severe atrial fibrosis;
3. Nonresponse or intolerance to ≥1 antiarrhythmic drug.

Exclusion Criteria:

1. With uncontrolled congestive heart failure;
2. Having significant valvular disease;
3. With myocardial infarction or stroke within 6 months of screening;
4. With Significant congenital heart disease;
5. Ejection fraction was <40% measured by echocardiography;
6. Allergic to contrast media;
7. Contraindication to anticoagulation medications;
8. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);
9. Left atrial (LA) thrombus;
10. Having any contraindication to right or left sided heart catheterization; 11. Previous atrial fibrillation ablation;

12. Presence of an implanted cardioverter-defibrillator; 13. Previous history of cardiac surgery; 14. Poor general health; 15. Life expectancy less than 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation (AF)/atrial flutter (AFL)/atrial tachycardia (AT) recurrence rate | up to 12 months after enrollment
  AF/AFL/AT recurrence is defined as presence of documented AF/AFL/AT episodes of 30 seconds or longer duration

SECONDARY OUTCOMES:
Postoperative AF recurrence rate | up to 12 months after enrollment
  AF recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration
Postoperative AFL/AT rate | up to 12 months after enrollment
  occurrence of AFL/AT is defined as presence of documented AFL/AT episodes of 30 seconds or longer duration
Incidence of complications | up to 12 months after enrollment
  death, atrioesophageal fistula, cardiac tamponade/perforation, myocardial infarction, stroke/cerebrovascular accident, thromboembolism, diaphragmatic paralysis, pneumothorax, pleural effusion, heart block, pulmonary vein stenosis, pulmonary edema, pericarditis and major vascular access complication or bleeding
Changes in the diameter of the left atrium and the left ventricular ejection fraction | up to 12 months after enrollment
  Changes in the diameter of the left atrium and the left ventricular ejection fraction